CLINICAL TRIAL: NCT02972541
Title: NeoAdjuvant Chemotherapy Versus Surgery Alone After Stent Placement for Left-sided Obstructive Colonic Cancer:a Multicenter, Controlled, Open-label Clinical Trial (NACSOC Trial)
Brief Title: Neoadjuvant Chemotherapy Verse Surgery Alone After Stent Placement for Obstructive Colonic Cancer
Acronym: NACSOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zhen Jun Wang, professor, Beijing Chao Yang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-161-1
Record Dates: First submitted 2016-09-08; First posted 2016-11-23 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer; Neoadjuvant Chemotherapy; Stent; Obstruction
MeSH Terms: conditions — Colorectal Neoplasms; Bites and Stings | interventions — Stents; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stenting with neoadjuvant chemotherapy (Experimental): After clinical success of colonic stenting, patients will receive neoadjuvant chemotherapy with mFOLFOX6 regimen for 3 cycles or CapeOx regimen for 2 cycles. Patients will undergo surgery 3-5 weeks after the last cycle of chemotherapy, type and extent of the surgery will be selected by the surgeon.
  Interventions: Device: Stenting with neoadjuvant chemotherapy
- Stenting with Immediate Surgery (Active Comparator): After clinical success of colonic stenting, patients will undergo surgery 7-14 days after inclusion. Type and extent of the elective surgery will be selected by the surgeon.
  Interventions: Device: Stenting with immediate Surgery

INTERVENTIONS:
Device: Stenting with neoadjuvant chemotherapy — After clinical success of colonic stenting, patients will be given neoadjuvant chemotherapy. Surgery is performed after 3 cycles of mFOLFOX6 or 2 cycles of CapeOx. The choice of surgery performed is up to the individual consultant colorectal surgeon. Patients will receive 5-9 cycles of mFOLFOX6 or 4-6 cycles of CapeoX after surgery. Each cycle of mFOLFOX6 consists of racemic leucovorin 400 mg/m², oxaliplatin 85 mg/m² in a 2-h infusion, bolus fluorouracil 400 mg/m² on day 1, and a 46-h infusion of fluorouracil 2400 mg/m². Each cycle of CapeOx consists of oxaliplatin 130 mg/m2, capecitabine 100 mg/m2 twice daily for 14 days.
  Arms: Stenting with neoadjuvant chemotherapy
Device: Stenting with immediate Surgery — After clinical success of colonic stenting, patients will undergo surgery 7-14 days later. The choice of surgery performed is up to the individual consultant colorectal surgeon. Patients will receive 8-12 cycles of mFOLFOX6 or 6-8 cycles of CapeoX after surgery. Each cycle of mFOLFOX6 consists of racemic leucovorin 400 mg/m², oxaliplatin 85 mg/m² in a 2-h infusion, bolus fluorouracil 400 mg/m² on day 1, and a 46-h infusion of fluorouracil 2400 mg/m². Each cycle of CapeOx consists of oxaliplatin 130 mg/m2, capecitabine 100 mg/m2 twice daily for 14 days.
  Arms: Stenting with Immediate Surgery

SUMMARY:
Colorectal cancer is the fourth most common cancer in China. Up to 30% of patients with colorectal cancer present with an emergency obstruction of the large bowel at the time of diagnosis, and 70% of all malignant obstruction occurs in the left-sided colon. Patients with obstruction are associated with worse oncologic outcomes compared with those having nonobstructive tumors. Conventionally, patients with malignant large bowel obstruction receive emergency surgery, with morbidity rates of 30%-60% and mortality rates of 7-22%, and about two-thirds of such patients end up with a permanent stoma.

Self-expanding metallic stents (SEMS) haven been used as a bridge to surgery (to relieve obstruction prior to elective surgery) in patients with potentially resectable colorectal cancer. Several clinical trials demonstrate that SEMS as a bridge to surgery may be superior to emergency surgery considering the short-term outcomes. SEMS is associated with lower morbidity and mortality rate, increased primary anastomosis rate, and decreased stoma creation rate. Although about half of patients can achieve primary anastomosis after stent placement, the primary anastomosis rate is still significantly lower compared with nonobstructing elective surgery. The interval between stent placement and surgery may be not long enough that bowel decompression is insufficient at the time of operation. Furthermore，the long-term oncologic results regarding SEMS as a bridge to surgery are still limited and contradictory. Sabbagh et al. suggest worse overall survival of patients with SEMS insertion compared with emergency surgery, the 5-year cancer-specific mortality was significantly higher in the SEMS group (48% vs 21%, respectively, P=0.02). One interpretation is that tumor cells may disseminate during the procedure of colonic stenting placement. We hypothesis that immediate chemotherapy after stenting may improve overall survival by eradicating micrometastasis. Moreover, neoadjuvant chemotherapy prolongs the interval between stent placement and surgery, and the time for bowel decompression is more sufficient, which may increase the success rate of primary anastomosis and decrease risk of stoma formation.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically proven colonic obstruction of the left colon/upper rectum presumed secondary to a carcinoma
* Able to give written, informed consent
* Primary tumor was resectable
* ECOG score 0 or 1
* Haemoglobin greater than 100 g/L after transfusion before chemotherapy,
* White blood cells greater than 3.0×10⁹ /L
* Platelets greater than 100×10⁹ / L;
* Glomerular filtration rate greater than 50 mL per minute as calculated by the Wright or Cockroft formula
* Bilirubin less than 1.5×Upper Limit of Normal(ULN)
* ALT and AST less than 2.5×ULN

Exclusion Criteria:

* Distal rectal cancers(equal or less than 10cm from the anal verge)
* Patients with signs of peritonitis and/or bowel perforation
* Patients who did not give informed consent
* Patients who were considered unfit for operative treatment or refuse surgery.
* Patients with suspected or proven metastatic adenocarcinoma;
* Patients with unresectable colorectal cancer, or planning for palliative treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2016-09-30; Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | From date of randomization until the date of tumor recurrence or death from any cause, assessed up to 5 years
Overall survival | From date of randomization until the date of death from any cause, assessed up to 5 years
Rate of stoma formation | From date of randomization until the follow-up ended, assessed up to 5 years

SECONDARY OUTCOMES:
Surgical complication | From date of randomization until the first follow-up ended, assessed up to 30 days
  Including but not limited to: anastomotic leakage, wound infection, intra-abdominal sepsis,perioperative mortality, etc.
Rates of primary colorectal anastomosis | From date of randomization until the first follow-up ended, assessed up to 30 days
  The primary colorectal anastomosis was defined as: the patients received one-stage surgery and colorectal anastomosis.
R0 resection rate | From date of randomization until the first follow-up ended, assessed up to 30 days
  R0 resection is defined as negative resection margins and no residual tumor.
Re-operation rate | From date of randomization until the follow-up ended, assessed up to 5 years
Chemotherapy complete rate | From date of randomization until the chemotherapy ended, assessed up to 1 years
Chemotherapy related complication | From date of randomization until the chemotherapy ended, assessed up to 1 years

CONTACTS AND LOCATIONS:
Overall Officials: zhenjun wang, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (32):
- China (32):
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Department of Colorectal Surgery, Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - the Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - the First Affiliated Hospital of Guangxi Medical University, Nanjing, Guangxi
  - Fourth Hospital of Hebei Medicial University, Shijiazhuang, Hebei
  - First Affiliated Hospital of Jiamusi University, Jiamusi, Heilongjiang
  - the 150th Central Hospital of Chinese PLA, Luoyang, Henan
  - the First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - the Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hubei General Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - the Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Provincial People'S Hospital, Changsha, Hunan
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - the First Affiliated Hospital of Dalian Medical University, Dalian, Shandong
  - Shandong Provincial Qianfoshan Hospital, Jinan, Shandong
  - Shandong General Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - the Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanxi Tumor Hospital, Taiyuan, Shanxi
  - the First Affiliated Hospital of Xi'An Jiaotong University, Xi’an, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - the First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Jinhua Hospital of Zhejiang University, Jinhua, Zhejiang
  - the Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sabbagh C, Browet F, Diouf M, Cosse C, Brehant O, Bartoli E, Mauvais F, Chauffert B, Dupas JL, Nguyen-Khac E, Regimbeau JM. Is stenting as "a bridge to surgery" an oncologically safe strategy for the management of acute, left-sided, malignant, colonic obstruction? A comparative study with a propensity score analysis. Ann Surg. 2013 Jul;258(1):107-15. doi: 10.1097/SLA.0b013e31827e30ce. PMID 23324856
- [Background] van Hooft JE, Bemelman WA, Oldenburg B, Marinelli AW, Lutke Holzik MF, Grubben MJ, Sprangers MA, Dijkgraaf MG, Fockens P; collaborative Dutch Stent-In study group. Colonic stenting versus emergency surgery for acute left-sided malignant colonic obstruction: a multicentre randomised trial. Lancet Oncol. 2011 Apr;12(4):344-52. doi: 10.1016/S1470-2045(11)70035-3. PMID 21398178
- [Background] Young CJ, De-Loyde KJ, Young JM, Solomon MJ, Chew EH, Byrne CM, Salkeld G, Faragher IG. Improving Quality of Life for People with Incurable Large-Bowel Obstruction: Randomized Control Trial of Colonic Stent Insertion. Dis Colon Rectum. 2015 Sep;58(9):838-49. doi: 10.1097/DCR.0000000000000431. PMID 26252845
- [Background] Huang X, Lv B, Zhang S, Meng L. Preoperative colonic stents versus emergency surgery for acute left-sided malignant colonic obstruction: a meta-analysis. J Gastrointest Surg. 2014 Mar;18(3):584-91. doi: 10.1007/s11605-013-2344-9. Epub 2013 Oct 30. PMID 24170606
- [Background] Ohman U. Prognosis in patients with obstructing colorectal carcinoma. Am J Surg. 1982 Jun;143(6):742-7. doi: 10.1016/0002-9610(82)90050-2. PMID 7046484
- [Background] Kim JS, Hur H, Min BS, Sohn SK, Cho CH, Kim NK. Oncologic outcomes of self-expanding metallic stent insertion as a bridge to surgery in the management of left-sided colon cancer obstruction: comparison with nonobstructing elective surgery. World J Surg. 2009 Jun;33(6):1281-6. doi: 10.1007/s00268-009-0007-5. PMID 19363580
- [Derived] Han J, Wang Z, Dai Y, Li X, Qian Q, Wang G, Wei G, Zeng W, Ma L, Zhao B, Wang Y, Yang K, Ding Z, Hu X. [Preliminary report on prospective, multicenter, open research of selective surgery after expandable stent combined with neoadjuvant chemotherapy in the treatment of obstructive left hemicolon cancer]. Zhonghua Wei Chang Wai Ke Za Zhi. 2018 Nov 25;21(11):1233-1239. Chinese. PMID 30506533